CLINICAL TRIAL: NCT02661529
Title: Enhancement of Contrast Opacification for Echocardiographic Imaging of the Right Heart and Shunts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Garvan C. Kane, M.D., Ph.D., M.D./Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 15-004591
Record Dates: First submitted 2015-09-29; First posted 2016-01-22 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Bidirectional Cardiovascular Shunt
Keywords: Shunt; Echocardiogram
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transesophageal Echocardiogram (Active Comparator): Patients undergoing an Transesophageal Echocardiogram (TEE) for diagnostic purposes to detect a cardiac shunt abnormality, using Saline/Air Mixture and Saline/Blood Mixture for vessel contrast
  Interventions: Procedure: Transesophageal Echocardiogram (TEE); Other: Saline/Air Mixture; Other: Saline/Blood Mixture
- Transthoracic Echocardiogram (Active Comparator): Patients undergoing an Transthoracic Echocardiogram (TTE) for diagnostic purposes to detect a cardiac shunt abnormality, using Saline/Air Mixture and Saline/Blood Mixture for vessel contrast
  Interventions: Procedure: Transthoracic Echocardiogram (TTE); Other: Saline/Air Mixture; Other: Saline/Blood Mixture

INTERVENTIONS:
Procedure: Transesophageal Echocardiogram (TEE) — Transesophageal echocardiography (TEE) is a test that produces pictures of the heart. TEE uses high-frequency sound waves (ultrasound) to make detailed pictures of the heart and the arteries that lead to and from it. Unlike a standard echocardiogram, the echo transducer that produces the sound waves for TEE is attached to a thin tube that passes through the mouth, down the throat and into the esophagus. Because the esophagus is so close to the upper chambers of the heart, very clear images of those heart structures and valves can be obtained.
  Arms: Transesophageal Echocardiogram
Procedure: Transthoracic Echocardiogram (TTE) — An echocardiogram is a type of ultrasound test that uses high-pitched sound waves that are sent through a device called a transducer. The device picks up echoes of the sound waves as they bounce off the different parts of the heart. These echoes are turned into moving pictures of the heart that can be seen on a video screen.
  Transthoracic echocardiogram (TTE) is the most common type of echocardiogram. Views of the heart are obtained by moving the transducer to different locations on the chest or abdominal wall.
  Arms: Transthoracic Echocardiogram
Other: Saline/Air Mixture — The Saline/Air mixture consists of 10 milliliters of sterile saline and 0.5 milliliters of air agitated together in a syringe prior to injection.
Other: Saline/Blood Mixture — The Saline/Blood mixture consists of 9 milliliters of sterile saline and 0.5 - 1.0 milliliters of blood agitated together in a syringe prior to injection.

SUMMARY:
The study aims to answer whether the use of a mixture of blood and saline alone (limited air) provides the same degree of right-heart contrast enhancement as compared to the standard agitated saline (with air), during two types of echocardiograms.

DETAILED DESCRIPTION:
A cardiovascular shunt is an abnormality of the blood flow between the sides of the heart or between the systemic and pulmonary circulation. A right-to-left shunt diverts blood from the right side of the heart to the left side or from the pulmonary to the systemic circulation through an anomalous opening such as septal defect or patent ductus arteriosus. To visualize the shunt during an echocardiogram, agitated saline solution is injected intravenously to provide air microbubble contrast which opacifies (makes visible) the right heart chambers and is the standard used for the non-invasive detection of right to left intracardiac or intrapulmonary shunts. However, agitated saline has the potential risk of air microembolism. Although this type of adverse event is uncommon (<1% of strokes are related to air embolism), there have been reports in the literature of a number of small strokes/transient ischemic attacks following agitated saline injections at the time of echocardiographic studies. Mixing blood with saline substantially reduces the amount of air introduced, and this study will attempt to quantify the differences in the degree of contrast enhancement.

100 patients scheduled for either Transesophageal Echocardiogram (TEE) or Transthoracic Echocardiogram (TTE) will be studied to determine the degree of contrast enhancement, when using a Saline/Air mixture versus a Saline/Blood mixture. Fifty participants of each type of echocardiography will be studied. The standard agitated saline mixture consists of 10 milliliters of sterile saline and 0.5 milliliters of air agitated together in a syringe prior to injection. The agitated Saline/Blood mixture consists of 9 milliliters of sterile saline and 0.5 - 1 milliliter of blood and agitated together in a syringe prior to injection.

All study participants will complete the routine clinical echocardiography (either a TEE or a TTE) with peripheral injection of agitated Saline/Air mixture, via an intravenous (IV) cannula attached to a three way stop cock. Blood removed from the patient will be withdrawn through the IV into a syringe and agitated with saline and then re-injected into the patient through the same tubing. After completion of the standard clinical imaging for shunt, the Saline/Blood mixture will be infused and an image obtained for comparison.

For each study, digital images will be stored and an Investigator who does not know which treatment arm/mixture was used for a given image, will subsequently rate image quality and assign an image score using a semi-quantitative scale: 0 = poor/no right atrial opacification, 1 = average right atrial opacification, 2 = good right atrial opacification. After all images are analyzed, the scores will be compared for both TEE and TTE studies.

ELIGIBILITY:
Inclusion Criteria

* Subjects having clinically indicated transesophageal or transthoracic echocardiogram, as ordered by their physician to detect a shunt.

Exclusion Criteria

* Unwillingness to provide consent to participate in the study

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Degree of right atrial opacification on echocardiogram image | Day 1
  The degree of right atrial opacification during echocardiogram will be rated with an image score; 0: poor/no opacification, 1: average opacification, 2: good opacification

CONTACTS AND LOCATIONS:
Overall Officials: Garvan Kane, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Ali MA, Hepinstall MJ, Cassidy CS, Lane CM, Pellikka PA, Thaden JJ, Pislaru SV, Kane GC. Agitated Blood-Saline Rather Than Agitated Air-Saline for Echocardiographic Shunt Studies. J Am Soc Echocardiogr. 2020 Aug;33(8):1032-1033. doi: 10.1016/j.echo.2020.03.014. Epub 2020 Jun 10. No abstract available. PMID 32532644